CLINICAL TRIAL: NCT02228486
Title: Alcohol Cue-Reactivity in Patients With Alcohol Dependency and Effects of Transcranial Direct Current Stimulation (tDCS) on Cue-exposure Therapy
Brief Title: Relapse Prevention in Alcohol Dependency by Transcranial Direct Current Stimulation Supported Cue Exposure Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Ann-Christine Ehlis, Dr., University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: aCR
Record Dates: First submitted 2014-08-15; First posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Alcohol Dependency
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cue Exposure Therapy and verum tDCS (Active Comparator): During alcohol cue exposure, an active tDCS with a duration of 15 minutes and 2 mA is applied to the left dorsolateral prefrontal cortex (F3, anode) and a reference electrode placed over Fp2 (electrode positions determined by the international 10-20 system). The electrodes are rectangular (35cm2).
  Interventions: Device: tDCS; Behavioral: Cue Exposure Therapy
- Cue Exposure Therapy and sham tDCS (Placebo Comparator): During alcohol cue exposure, a placebo tDCS is used with electrodes placed over the left dorsolateral prefrontal cortex (F3, anode) and a reference electrode placed over Fp2 (electrode positions determined by the international 10-20 system). The electrodes are rectangular (35cm2). There is a 20 second ramp going up until 2 mA and back to 0 again at the beginning and the end of the placebo stimulation with no active stimulation during the cue exposure.
  Interventions: Behavioral: Cue Exposure Therapy
- Waiting list control group (No Intervention): The Cue-Reactivity of patients assigned to this arm will be measured twice with an interval of 5 weeks. Afterwards, patients will take part in the cue exposure therapy like subjects assigned to the active arms of the study

INTERVENTIONS:
Device: tDCS — 2 mA (verum group) over the left dorsolateral prefrontal cortex (F3, anodal), 15 min; 10 seconds ramp in verum and sham group (see also above)
  Other Names: transcrancial direct currenct stimulation
  Arms: Cue Exposure Therapy and verum tDCS
Behavioral: Cue Exposure Therapy — 5 weeks (9 sessions) of cue-exposure therapy with preferred alcoholic beverage (see also above)
  Other Names: Cue-Exposure Training
  Arms: Cue Exposure Therapy and sham tDCS; Cue Exposure Therapy and verum tDCS

SUMMARY:
Relapse is a major risk in substance abuse disorders, which is closely related to craving for a substance, describing a strong urge for consumption. Cue-exposure therapy is an intervention aiming at the reduction of perceived craving by repeated confrontation. It is based on the assumption that craving drops after repeated exposure without the reinforcing experience elicited by consumption. In the present study, patients with alcohol dependency take part in nine cue-exposure training sessions. Each session consists of mood induction reflecting a high risk situation with subsequent in vivo confrontation with one's preferred alcoholic beverage followed by the training of coping strategies. During the cue-exposure, patients focus on perceiving automatic responses to alcohol-related cues. We hypothesize that especially patients exhibiting initially high reactions to such cues should profit from this intervention the most. The reactions are measured on a subjective (craving) and physiological level (hemodynamics of the prefrontal cortex, heart rate variability, electrodermal activity). Furthermore, we want to strengthen the expected training effects during the cue-exposure by an activating transcranial direct current stimulation of the dorsolateral prefrontal cortex, which has been shown to be hypoactive in substance abuse disorders. We investigate how the cue-exposure training affects the processing of alcoholic cues (cue-reactivity) and its relation to clinical symptoms of alcohol dependency.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of an alcohol dependence (F10.2)
* abstinence motivation

Exclusion Criteria:

* epileptic seizures
* acute psychotic episode
* another substance use disorder besides nicotine dependency (F17.2)
* acute withdrawal symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
alcohol consumption days | six months

SECONDARY OUTCOMES:
Maximum subjective alcohol craving during alcohol cue-exposure (10-point scale) | 5 weeks
  During alcohol cue-exposure, subjects rate the subjective craving regularly on a scale from 0 to 10.
subjective rating of self-efficacy (score on a 10 item-scale) | 6 months
  questionnaire (General Self-Efficacy Scale, Schwarzer & Jerusalem, 1995)

OTHER OUTCOMES:
Hemodynamics in the orbitofrontal cortex and the dorsolateral prefrontal cortex during cue-exposure | 5 weeks
  With near-infrared spectroscopy, changes in the concentrations of oxygenated (O2HB) and deoxygenated (HHb) haemoglobin are assessed (in mmol*mm), peaks in those concentrations are evaluated
heart-rate variability during alcohol cue-exposure | 5 weeks
  low frequency/ high frequency (LF/HF) power ratio and standard deviation of the duration between R-peaks (RR) during cue-exposure
Skin conductance level during alcohol cue exposure | 5 weeks
  skin conductance level (SCL) in Mikrosiemens (μS)

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Christine Ehlis, PhD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- Department of Psychiatry and Psychotherapy, University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany